CLINICAL TRIAL: NCT05462665
Title: Evaluation of the Intravenous Tissue Plasminogen Activator Treatment Algorithm of Nursing Intern Students and Evaluation of the Efficiency of Simulation Method in the Development of Self-Efficacy Proficiency Levels
Brief Title: Evaluation of the Intravenous Tissue Plasminogen Activator Treatment Algorithm of Nursing Intern Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, OZGE SOYDANER, nurse, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: tPA Treatment
Record Dates: First submitted 2022-03-23; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2021-12

CONDITIONS: Acute Stroke
Keywords: tissue plasminogen activator; acute stroke; intravenous tissue plasminogen activator; nursing care; neurology nursing; acute stroke treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intern nurses will be numbered from 1 to 75 and will be randomly divided into study and control groups from the random numbers table.
  After the groups are determined by the randomization method, each intern nurse in the study and control groups will be interviewed face to face and their written informed consent will be obtained. Then, all nursing intern students participating in the research will be asked to fill in the IV tPA Treatment Knowledge Level Evaluation Form, Self-Efficacy Competence Scale. Intern nurses in both groups will be given 1-hour theoretical training on IV tPA treatment before, during and after the procedure. In addition, simulation-based training will be applied to the intern nurses in the study group regarding IV tPA treatment before, during and after the procedure.
Who Masked: Participant
Masking Description: Intern nurses will be numbered from 1 to 75 and will be randomly divided into study and control groups from the random numbers table.
  After the groups are determined by the randomization method, each intern nurse in the study and control groups will be interviewed face to face and their written informed consent will be obtained. Then, all nursing intern students participating in the research will be asked to fill in the IV tPA Treatment Knowledge Level Evaluation Form, Self-Efficacy Competence Scale. Intern nurses in both groups will be given 1-hour theoretical training on IV tPA treatment before, during and after the procedure. In addition, simulation-based training will be applied to the intern nurses in the study group regarding IV tPA treatment before, during and after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Nursing intern students (n:39) will be given theory training about tPA treatment
  Interventions: Behavioral: theory training
- Control (Experimental): Nursing intern students (n:39) will be given theory training and simulation training about tPA treatment
  Interventions: Behavioral: theory training; Behavioral: theory and simulation training

INTERVENTIONS:
Behavioral: theory training — theory training
  Other Names: tPA treatment knowledge of nursing students will increase
Behavioral: theory and simulation training — theory and simulation training
  Other Names: tPA treatment knowledge of nursing students will increase
  Arms: Control

SUMMARY:
Intravenous (IV) tissue plasminogen activator (tPA) is one of the key elements of acute ischemic stroke. In this study, acute stroke patients maximum benefit from the treatment, intravenous tissue plasminogen activator (IV tPA) minimizing the errors related to the treatment of acute ischemic stroke patients of nursing students from clinical practice guides published on the treatment of It is aimed to be informed and to standardize nursing interventions.

DETAILED DESCRIPTION:
Time management in acute stroke patients is possible with a multidisciplinary approach and team members who have received specific training for acute stroke patients. Studies have shown that the maximum result of treatment for acute stroke patients depends on nurses' ability to identify disease symptoms, plan and apply symptom-specific nursing care. There is evidence that the multidisciplinary presence of stroke teams in stroke units and the delivery of coordinated care during the acute phase improve patient outcomes . Coordinated care by the stroke team improves patient outcomes, reduces hospital costs, reduces patient readmission, and improves patient care quality.

ELIGIBILITY:
Inclusion Criteria:

Intern nursing student at Dokuz Eylül University

Exclusion Criteria:

Those who did not agree to participate in the study Those who were not be intern

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
self-efficacy scale | Change from baseline in Intravenous Tissue Plasminogen Activator Treatment knowledge and 2 weeks after intervention
  Effectiveness change of Intravenous tissue plasminogen activator treatment knowledge after theoric teaching
simulation scale | 2 weeks after simulation training
  evaluation the simulation design
tPA treatment information form | Change from baseline in Intravenous Tissue Plasminogen Activator Treatment knowledge and 2 weeks after intervention
  Effectiveness change of Intravenous tissue plasminogen activator treatment knowledge after simulation and theoric teaching

CONTACTS AND LOCATIONS:
Overall Officials: GULSAH GUROL ARSLAN, Study Director — DOKUZ EU
Locations (1):
- Ozge Soydaner, Izmir, Turkey (Türkiye)